CLINICAL TRIAL: NCT02781246
Title: Effect of Perineural Dexmedetomidine on the ED50 Ropivacaine for Brachial Plexus Blocks in Pediatric Patients: a Randomized Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Wenhua Zhang, Director, Clinical Resesearch, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Wzhang05
Record Dates: First submitted 2016-05-16; First posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Dose-Response Relationship, Drug

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- saline (Group A) (Active Comparator): perineural ropivacaine
  Interventions: Drug: perineural dexmedetomidine
- 0.5 mcg/kg dexmedetomidine (Group B) (Active Comparator): (perineural ropivacaine plus 0.5 mcg/kg dexmedetomidine),
  Interventions: Drug: perineural dexmedetomidine
- 1 mcg/kg dexmedetomidine (Group C) (Active Comparator): (perineural ropivacaine plus 1 mcg/kg dexmedetomidine)
  Interventions: Drug: perineural dexmedetomidine
- 1.5 mcg/kg dexmedetomidine (Group D) (Active Comparator): (perineural ropivacaine plus 1.5mcg/kg dexmedetomidine)
  Interventions: Drug: perineural dexmedetomidine
- 2 mcg/kg dexmedetomidine (Group E) (Active Comparator): (perineural ropivacaine plus 2 mcg/kg dexmedetomidine)
  Interventions: Drug: perineural dexmedetomidine

INTERVENTIONS:
Drug: perineural dexmedetomidine — Children scheduled for arm and forearm surgery underwent supraclavicle brachial plexus blocks with ropivacaine and dexmedetomidine guided by ultrasound visualisation were randomly assigned five groups: Group A (perineural ropivacaine), Group B (ropivacaine plus 0.5 mcg/kg dexmedetomidine), Group C (ropivacaine plus 1 mcg/kg dexmedetomidine), Group D (ropivacaine plus 1.5mcg/kg dexmedetomidine) and Group E (ropivacaine plus 2 mcg/kg dexmedetomidine). In each group, children received a certain concentration of ropivacaine which adjusted by the "Dixon up-and-down method for supraclavicle brachial plexus. The first child received 0.2% ropivacaine , and the concentration of ropivacaine varied by 0.1% according to the up-and-down method. The primary endpoint was the minimum local anesthetic concentration (MLAC).

SUMMARY:
Dexmedetomidine can prolong the duration of local anesthetics, but the effect of perineural dexmedetomidine on the potency of ropivacaine for brachial plexus blocks in pediatric patients has not been investigated. This study was designed to determine the effect of perineural dexmedetomidine on ropivacaine for brachial plexus blocks in pediatric patients

DETAILED DESCRIPTION:
150 children scheduled for arm and forearm surgery underwent supraclavicle brachial plexus blocks with ropivacaine guided by ultrasound visualisation were randomly assigned to one of the five groups: Group A (perineural ropivacaine), Group B (ropivacaine plus 0.5 mcg/kg dexmedetomidine), Group C (ropivacaine plus 1 mcg/kg dexmedetomidine), Group D (ropivacaine plus 1.5mcg/kg dexmedetomidine) and Group E (ropivacaine plus 2 mcg/kg dexmedetomidine). The primary endpoint was the minimum local anesthetic concentration (MLAC), which was determined using the Dixon up-and-down method. The secondary endpoints were the duration of analgesia and sedation

ELIGIBILITY:
Inclusion Criteria:

* ASA I,II children, aged between 2 and 6 years, who were scheduled for arm and forearm surgery underwent supraclavicular brachial plexus blocks.

Exclusion Criteria:

* any subjects with neurological, neuromuscular, psychiatric, or blood clotting disorders, or known history of active and severe renal, hepatic, respiratory, or cardiac diseases, or known allergy to systemic or local anesthetics or dexmedetomidine

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the minimum local anesthetic concentration (MLAC) | up to 30 minutes after brachial plexus blocks
  For each patient, the target concentration of perineural ropivacaine was determined using the modified Dixon's up-and-down method starting with 0.20% in each group, varied with 0.1% as a step size. Increasing or decreasing the target concentration of perineural ropivacaine was determined by the response of the previous child in the same group. The response of each child was observed for 60 s after the skin incision and evaluated as 'successful' or 'unsuccessful.' 'Unsuccessful' was recorded when skin incision caused motor responses or change in hemodynamic parameters (heart rate and mean blood pressure) more than 20% of the preincision values. If the response was determined to be unsuccessful, the concentration of perineural ropivacaine given to the next patient would be increased by 0.1%. If it was successful, the concentration of caudal levobupivacaine given to the next patient would be decreased by 0.1%
Postoperative pain | up to 12 hours after brachial plexus blocks
  The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain.
  The scale is scored in a range of 0-10 with 0 representing no pain, 1-3 representing mild uncomfortable, 4-6 representing moderate pain, 7-10 representing high-level pain or/and uncomfort. The FLACC scale was evaluated at 6 and 12 hours postoperatively, and scale of ≥4 points was regarded as an inadequate analgesia and was managed with 10 mg/kg of ibuprofen by mouth every 6 h as required
The sedation status | up to 12 hours after brachial plexus blocks
  Sedation status was evaluated by a attending anesthesiologists with a 6-point sedation scale, which was modified from the Modified Observer Assessment of Alertness and Sedation Scale (MOAA/S). The MOAA/S scale was evaluated at 6 and 12 hours postoperatively
  0 Does not respond to a noxious stimulus
  1. Does not respond to mild prodding or shaking
  2. Responds only after mild prodding or shaking
  3. Responds only after name is called loudly or repeatedly
  4. Lethargic response to name-spoken in normal tone
  5. Appears asleep, but responds readily to name-spoken in normal tone
  6. Appears alert and awake, responds readily to name-spoken in normal tone

SECONDARY OUTCOMES:
pulse oximetry | up to 12 hours after brachial plexus blocks
  Significant Oxyhemoglobin desaturation was defined as < 90%
heart rate | up to 12 hours after brachial plexus blocks
  Bradycardia was defined as a reduction in heart rate more than 20% from the baseline values
noninvasive arterial blood pressure | up to 12 hours after brachial plexus blocks
  Hypotension was defined as a reduction in systolic blood pressure more than 20% from the baseline values